CLINICAL TRIAL: NCT06585137
Title: Effect of a Web-Based Mind-Body Awareness Program Based on Meleis Transition Theory on Women Receiving Infertility Treatment: A Randomized Controlled Study
Brief Title: Impact of a Web-Based Mind-Body Awareness Program on Women Undergoing Infertility Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: Assistant Professor Onur İNCE (Unknown); Associate Professor Dr. Çiğdem YÜCEL ÖZÇIRPAN (Unknown)
Responsible Party: Principal Investigator, Gülşah VURAL AKTAN, Nurse, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PhD-01
Record Dates: First submitted 2024-08-28; First posted 2024-09-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Infertility, Female
Keywords: Nursing; Infertility; Nursing Theory; Fertility; Awareness; Meleis; Fertility readiness
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based mind-body awareness program (Active Comparator): Participants in the intervention group will participate in a web-based mind-body awareness program.
  Interventions: Other: Web-Based Mind-Body Awareness Program
- Routine nursing care (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Web-Based Mind-Body Awareness Program — The program has been developed in line with peer-reviewed literature and expert opinions. It will incorporate a nursing approach based on the Meleis transition theory, education, mind-body awareness practices, and messages specific to women's health. Participants will be involved in an awareness program consisting of 3 sessions over an average of 2 weeks. Participants will be asked to complete their first final test one day after the egg retrieval (OPU) procedure, i.e., an average of 8-12 days after ovulation induction. There will be no intervention between the embryo transfer and the pregnancy test day. During this time period, interactive sessions between the researcher and participants will be conducted, and nursing care will be provided according to Meleis. The implementation phase of the study will be completed with 39 participants after the second final test following the pregnancy test.
  Arms: Web-based mind-body awareness program

SUMMARY:
The goal of this two-group parallel randomized controlled study is to determine the effect of a web-based mind-body-based awareness program based on Meleis Transition Theory on fertility awareness and readiness levels in women receiving infertility treatment.

DETAILED DESCRIPTION:
Developing fertility awareness in women receiving infertility treatment can enable changes in lifestyle habits that can increase fertility. Having and increasing fertility awareness in infertile individuals can increase the likelihood of pregnancy and having a healthy pregnancy, positively affect general health and reproductive health, and change negative lifestyle habits that can affect the treatment process for infertility. Fertility readiness can be provided with fertility awareness and can positively affect treatment outcomes. This research will be conducted as a two-group parallel randomized controlled trial to determine the effect of a web-based mind-body awareness program based on Meleis Transition Theory on fertility awareness and readiness levels in women receiving infertility treatment. The research will be conducted with women receiving infertility treatment at the In Vitro Fertilization Unit of Hacettepe University Faculty of Medicine. The sample will include women who volunteer to participate in the study, have started the infertility treatment process, have had at most two IVF attempts, speak and understand Turkish, are at least primary school graduates, are not in any psychological or social support group, have not completed or are not currently participating in any mind/body program for fertility. A total of 78 women will be included in the study sample: 39 for the intervention group and 39 for the control group. The Introductory Information Form, Fertility Awareness Scale, Fertility Readiness Scale, and Satisfaction Evaluation Form will be used to collect the data. Within the scope of the study, a web-based mind-body awareness program based on Meleis transition theory will be applied to the women in the intervention group. The routine nursing care in the unit will be applied to the control group. Research data will be analyzed using mean, standard deviation, median, quarts, percentage, minimum and maximum values, Chi-square, and Mann Whitney-U tests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Being diagnosed with primary infertility
* Starting the infertility treatment process
* Having attempted IVF at most twice before
* Being able to speak and understand Turkish
* Being at least a primary school graduate
* Not taking part in any psychological or social support group.
* Not having completed or currently participating in any mind/body program for fertility.

Exclusion Criteria:

* Women applying for frozen embryo transfer without ovarian stimulation
* Being diagnosed with secondary infertility
* Having a diagnosis of a chronic disease
* Having communication problems (vision, hearing)

Ages: 23 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-22 (Estimated)

PRIMARY OUTCOMES:
Fertility Awareness Scale | A pre-test will be administered before the study begins. Then, a post-test will be administered three times, 1 day after the OPU procedure, then at 3 months and 6 months.
  This scale was developed to measure fertility awareness in women. The scale is Likert-type and has 19 items and two sub-dimensions (Body Awareness, Cognitive Awareness). Items in the scale are scored from 1 to 5 (1-Never, 2-Rarely, 3-Occasionally, 4-Most of the time and 5-Always) and there are no reverse-scored items. Possible scores in total for the scale are 19-95, 10-50 for the "Body Awareness" sub-dimension, and 9-45 for the "Cognitive Awareness" sub-dimension. If the total score is between 19-43, the awareness level is interpreted as ''low'', if it is between 44-69, it is ''medium'', and if it is between 70-95, it is interpreted as ''high''.
Fertility Preparedness Scale for Women Receiving Fertility Treatment | A pre-test will be administered before the study begins. Then, a post-test will be administered three times, 1 day after the OPU procedure, then at 3 months and 6 months.
  The scale, consisting of 23 questions, was created to measure the readiness of women preparing to become pregnant. The scale consists of 3 sub-dimensions: "hope and awareness", "relaxed body and brain" and "positive feelings and thoughts". Since the scale items consist only of positive expressions, the scores obtained are calculated as they are. The scores of the items are 5, 4, 3, 2, and 1, respectively. The minimum score is 23, the maximum score is 115 on the scale, and a high score indicates that fertility preparedness is strong. The median score on the scale is 56. A score of 56 or higher on the scale indicates that the woman feels more prepared for pregnancy, while a lower score indicates that she feels less prepared.

SECONDARY OUTCOMES:
Introductory Information Form | FSH and E2 levels will be monitored on the 2nd-3rd day of the menstrual cycle, the number of oocytes collected on the 16th day of the cycle, embryo transfer status on the 18th day of the cycle, and pregnancy test on the 28th day of the cycle.
  Follicle-stimulating hormone (FSH) and estradiol (E2) levels, number of oocytes collected, embryo transfer status, and blood pregnancy test results will be taken from the patient file and added to the form.

CONTACTS AND LOCATIONS:
Overall Officials: Onur İNCE, MD, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Samanpazarı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No